CLINICAL TRIAL: NCT00976924
Title: Clinical Test of Blood Glucose Test Strips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andon Medical Co.,Ltd (Industry)
Responsible Party: Yi Liu, Andon Medical Co.,Ltd
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AndonMedical1
Record Dates: First submitted 2009-09-08; First posted 2009-09-15 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes
Keywords: blood glucose
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Andon (Experimental): Andon blood glucose test strips with test meter
  Interventions: Device: blood glucose monitor
- Lifescan (Active Comparator): Lifescan blood glucose test strips with test meter
  Interventions: Device: blood glucose monitor

INTERVENTIONS:
Device: blood glucose monitor — Blood glucose monitor is used to monitor the blood glucose level of the human-being.
  Other Names: Andon or lifescan blood glucose monitor

SUMMARY:
Blood glucose test strips are tested with the test meters to test the accuracy of the blood pressure monitoring function.

ELIGIBILITY:
Inclusion Criteria:

* The patients with blood glucose within the range of ISO15197

Exclusion Criteria:

* The patients with blood glucose out of the range of ISO15197

Ages: 22 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
blood glucose value | 5 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University general hospital, Tianjin, Tianjin Municipality, China